CLINICAL TRIAL: NCT02253524
Title: Comparison of Efficacy Dimenhydrinate and Metoclopramide in the Treatment of Nausea Due to Vertigo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bulent Erdur, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PAU-1179
Record Dates: First submitted 2014-09-09; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Nausea; Vomiting; Vertigo
Keywords: Metoclopramide; Dimenhydrinate; emergency medicine
MeSH Terms: conditions — Nausea; Vomiting; Vertigo | interventions — Dimenhydrinate; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dimenhydrinate (Active Comparator): 50 mg Dimenhydrinate with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes
  Interventions: Drug: Dimenhydrinate
- Metoclopramide (Active Comparator): 10 mg Metoclopramide with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Dimenhydrinate — 50 mg Dramamine with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes
  Other Names: Dramamine
  Arms: Dimenhydrinate
Drug: Metoclopramide — 10 mg Metoclopramide with 5 cc syringe in 150 ml normal saline given as a slow intravenous infusion over 15 minutes
  Other Names: Primperan; metpamid
  Arms: Metoclopramide

SUMMARY:
* Vertigo complaint is one of the common cause of patients who applied to emergency services.
* Patients who have applied to emergency services with vertigo complaint mostly have nausea as an additionally symptom to this complaint and anti-emetic agents can be used in their treatments very often.
* The investigators purpose is to investigate the advantages of Dimenhydrinate and metoclopramide to each other in the treatment of vertigo and the vertigo accompanied by nausea

DETAILED DESCRIPTION:
* Vertigo describes the illusion of being subject to an involuntary movement, usually rotational, of the patient or the patient's surroundings which is caused by sudden tonic neural activity.
* The management and episodic treatment of patients with spontaneous vertigo related nausea-vomiting symptoms are somewhat controversial in the emergency department setting.
* Patients admitted to the emergency department with complaints of vertigo in addition to a large portion of the symptoms are accompanied by nausea and antiemetic agents are frequently used in the treatment.
* An ideal treatment should be rapid in onset and effective, and lack debilitating side effects.
* Although a wide variety of classes of pharmacologic agents and modalities are used, the emergency department treatment of acute spontaneous vertigo and associated with nausea- vomiting has not been well studied.
* It has been reported that the most commonly used medications for parenteral treatment of vertigo and nausea-vomiting in emergency department are dimenhydrinate (DMT) and metoclopramide (MTP).
* It has a depressant action on hyper-stimulated labyrinthine function and antiemetic effects, believed to be due to the antihistamine.
* Dimenhydrinate inhibits vomiting by affecting the histaminic receptor and cholinergic receptor function center of vestibular nucleus in the central vestibular system.
* Dimenhydrinate reduces the symptoms of vertigo with depressant effects on the labyrinth function by this means.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 65 years old patients,
* had vertigo and accompanied nausea or vomiting [VAS (visual analog scale) score >5] during their emergency department episode of care for which the attending physician recommended intravenous antiemetic medication.

Exclusion Criteria:

* abnormal vital signs,
* women who were pregnant or lactation,
* those with a history of epilepsy,
* acute psychiatric symptoms,
* organic brain disease,
* parkinson's disease or phaeochromocytoma,
* or any known allergy to the study drugs,
* uncooperative individuals,
* use of any antiemetic drug in the previous 8 hours or previous delivery of intravenous fluids during the emergency department episode of care,
* currently undergoing chemotherapy or radiotherapy,
* mechanical obstruction or perforation,
* gastrointestinal bleeding,
* inability to understand study explanation or outcome measures (any reason),
* known allergy or previous adverse reaction to metoclopramide or dimenhydrinate,
* and patients who refused to participate study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
compare the effects of intravenous dimenhydrinate and metoclopramide in the treatment of nausea due to vertigo in emergency setting. (nausea and vertigo scores as measured by Visual Analogue Scale.) | Change from Baseline in nausea and vertigo scores at 30 minutes.
  - participants will be followed for the duration of hospital stay, an expected average of 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent ERDUR, proffessor, Study Director — Pamukkale University